CLINICAL TRIAL: NCT06929442
Title: A Randomized Controlled Trial of a Preventive Behavioral Intervention for Young Adults With Psychotic Experiences
Brief Title: A Preventive Behavioral Intervention for Young Adults With Psychotic Experiences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016P0023511
Record Dates: First submitted 2025-04-04; First posted 2025-04-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Psychotic Disorders; Mood Disorders; Anxiety Disorders
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized trial with active control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resilience Training (RT) (Experimental): RT is a 4-week program of weekly 90-minute sessions in which participants are taught the following skills: mindfulness, self-compassion and mentalization.
  Interventions: Behavioral: Resilience Training (RT)
- Life Skills Training (LST) (Active Comparator): LST is a 4-week program of weekly 90-minute sessions, in which participants are provided information about helpful life skills, including financial literacy, health, physical and internet safety.
  Interventions: Behavioral: Life Skills Training (LST)

INTERVENTIONS:
Behavioral: Resilience Training (RT) — RT is a 4-week program of weekly 90-minute sessions in which participants are taught the following skills: mindfulness, self-compassion and mentalization.
  Arms: Resilience Training (RT)
Behavioral: Life Skills Training (LST) — LST is a 4-week program of weekly 90-minute sessions, in which participants are provided information about helpful life skills, including financial literacy, health, physical and internet safety.
  Arms: Life Skills Training (LST)

SUMMARY:
This is a randomized controlled trial testing the efficacy of Resilience Training in college students with elevated transdiagnostic risk for developing a serious mental illness.

ELIGIBILITY:
Inclusion criteria:

1. 18-30 years old
2. Enrolled as a first or second year student (i.e., freshman or sophomore) in an undergraduate program at the college or university where the intervention takes place
3. Students who endorse some psychotic experiences (Peter's et al. Delusion Inventory (PDI) score > 3)

Exclusion criteria:

1. Inability to provide informed consent
2. Not proficient in English
3. Current self-reported Diagnostic Statistical Manual 5 (DSM-5) diagnosis with active symptoms (such as active psychotic symptoms, current suicidality, serious active alcohol or substance use, marked deterioration in functioning over the prior month) determined by clinical interview with participant, or self-report of a psychiatric diagnosis that necessitates close monitoring or individual therapy and/or inpatient or partial hospitalization
4. Current enrollment in psychological or behavioral health treatment.
5. Current use of psychotropic medications (other than stimulants) prescribed by a physician.
6. A diagnosis of a serious, chronic mental illness as determined by the Mini-International Neuropsychiatric Interview (MINI)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Peters Delusions Inventory | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Peters Delusions Inventory (PDI) is a brief 21-item survey using non-stigmatizing and non-clinical language that obtains ratings of common delusional experiences (e.g. paranoia, grandiosity, ideas of reference) and perceptual aberrations (e.g. experiences of being controlled; thought insertion, withdrawal, and echoing), i.e., psychotic experiences. The PDI also measures conviction, preoccupation, and distress related to these experiences. This scale is scored from 0-21, with higher scores indicating a greater number of experiences endorsed.

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Beck Depression Inventory (BDI) is a 21-item self-report assessment of symptoms of depression on a Likert scale of 0-63, with higher scores indicating more depressive symptoms.
Spielberger State-Trait Anxiety Inventory | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 20-item self-report scale measuring symptoms of anxiety, both those that are trait-like and ongoing, and those that are state-like and current. Scores range from 0-120, with higher scores indicate higher levels of anxiety symptoms.
Columbia-Suicide Severity Rating Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is an interview-based measure to identify and assess suicidal thoughts, behaviors and suicide risk. The interview consists of two subscales, an ideation and behavior subscale. The severity of ideation subscale is rated on a 5-point ordinal scale, with higher scores indicating a more detailed plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
UCLA Loneliness Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The UCLA Loneliness Scale is a 20-item scale to measure subjective feelings associated with loneliness. Scores range from 20 - 80, with higher scores indicating stronger degree of loneliness reported.
Temporal Experience of Pleasure Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Temporal Experience of Pleasure Scale (TEPS) is an 18-item questionnaire used to assess experiences of both anticipatory and consummatory aspects of pleasure. The Anticipatory score ranges from 10 - 60, with higher scores indicating greater pleasure. The Consummatory score ranges from 8 - 48, with higher scores indicating greater pleasure.
Anticipatory and Consummatory Interpersonal Pleasure Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) is a 17-item measure of both anticipatory and consummatory social pleasure. Scores range from 17 - 102, with lower equals indicating greater social anhedonia. The Anticipatory scale is scored between 10 - 60, wither higher scores indicating more pleasure. The Consummatory scale is scored from 7 - 42, with higher scores indicating more pleasure.
Time Alone Questionnaire | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Time Alone Questionnaire (TAQ) is a 6-item questionnaire used to assess the portion of waking hours spent with others, compared to the desired amount of time spent with others. Participants are asked to estimate the average percentage of their waking hours actually spent with other people versus alone (ranging from 0 - 1), and the percentage of their waking hours that they would prefer to spend with other people versus alone (ranging from 0 - 1).
Social Discomfort Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Social Discomfort Scale (SDS) is a 3-item questionnaire assessing to what extent - and reason for why - individuals are uncomfortable in the physical presence of others. Scores range from 1 - 6, with higher scores indicating higher levels of social discomfort.
Prodromal Questionnaire - Brief | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Prodromal Questionnaire - Brief (PQ-B) is a 9-item scale designed to assess subclinical symptoms of psychosis. Scores range from 0 - 21, with higher scores indicating more severe symptoms reported.
Phalen et al. Screener | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Phalen et al. Screener is a 4-item questionnaire used to assess subclinical psychotic symptoms (psychotic experiences). Scores range from 0 - 4, with higher scores indicating the presence of more psychotic symptoms.
Launay-Slade Hallucination Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Launay-Slade Hallucination Scale (LSHS) is a 16-item questionnaire used to assess hallucinatory experiences. Scores range from 0 - 64, with higher scores indicating greater frequency of hallucinations reported.
Structured Interview for Psychosis/Scale for the Assessment of Prodromal Symptoms | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Structured Interview for Psychosis/Scale for the Assessment of Prodromal Symptoms (SIPS/SOPS) is a measure of subclinical symptoms of psychosis. It is organized into four primary symptom sections, with a total of 19 items each rated on a scale from 0-6, with higher scores indicating higher symptom severity.
Connor-Davidson Resilience Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Connor-Davidson Resilience Scale (CD-RISC) is a 25-item self-report scale assessing levels of coping and emotional resilience. It is rated on a scale of 0-100, with higher scores indicating greater coping skills and emotional resilience.
Five Facet Mindfulness Questionnaire | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report survey assessing one's capacity for mindfulness. It contains 5 sub-scales. It is scored on a 0-195 scale, with higher scores indicating a greater capacity for mindfulness.
Self-Compassion Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Self-Compassion Scale (SCS) a 26-item scale for the assessment of self-compassion. Scores range from 16 - 80, with higher scores indicating better self-compassion reported.
Reflective Functioning Questionnaire | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  Reflective Functioning Questionnaire (RFQ) is a 31-item questionnaire to assess impairments in mentalization. Scores range from 31 - 217, with higher scores indicating better reflective functioning reported.
Positive and Negative Affect Schedule | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Positive and Negative Affect Schedule (PANAS) is a 20-item questionnaire for assessing positive and negative affect. It is organized into two primary sections, each section with 10 items, ranging from 1 - 5, with higher scores indicating stronger affect.
General Self-Efficacy Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The General Self-Efficacy Scale (GSE), is a 10-item questionnaire for the assessment of self-efficacy, the ability to cope with stressors. Scores range from 10 - 40, with higher scores indicating stronger self-efficacy reported.
Emotional Reactivity Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Emotional Reactivity Scale (ERS) is a 21-item self-report measure of emotional reactivity, comprised of emotion sensitivity, intensity, and persistence. Scores range from 0 - 44, with higher scores indicating greater emotional reactivity.
Difficulties in Emotion Regulation Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item questionnaire to assess how people regulate their emotions. Scores range from 36 - 180, with higher scores indicating greater impairment and difficulties in regulating emotions.
Perceived Stress Scale | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Perceived Stress Scale (PSS) is a 10-item, widely-used psychological instrument for measuring the perception of stress. Scores range from 0 - 40, with higher scores indicating greater perceived stress.
Emotion Recognition Task | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Emotion Recognition Task (ER40) assesses facial emotion recognition ability and includes 40 color photographs of faces. Recognition task accuracy percentage ranges from 0 - 1 (average over all 40 trials).
Emotion Differentiation Task | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Emotion Differentiation Task is a task with 36 face pairs (13 happy, 13 sad) measuring the ability to detect subtle differences in intensity within emotions. Differentiation task accuracy percentage ranges from 0 - 1 (average over all 36 trials).
Reading the Mind in the Eyes | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  Reading the Mind in the Eyes is an objective measure of Theory-of-Mind capacity, particularly the ability to read emotion.
Stop Distance Paradigm | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Stop Distance Paradigm is an objective measure for assessing the size and permeability of personal space.
Hippocampal-frontal functional connectivity | Baseline, 4-weeks, and 12 months
  The hippocampal-frontal functional connectivity measure is derived from functional magnetic resonance imaging (fMRI) data acquired during a 10 minute period when the participant is in a state of wakefulness but has no directed task. In the analyses, fluctuations in hippocampal activity during this period are correlated with activity fluctuations of frontal cortical regions to produce a measure of connectivity strength.
Fear conditioning responses of the hippocampus | Baseline, 4-weeks, and 12 months
  This measure is derived from fMRI data acquired when the participant is presented with faces, some of which have been associated with an aversive stimulus. In the analysis, hippocampal activation during blocks of non-aversive and aversive stimulus presentations are directly contrasted to produce a measure of fear conditioning activation.
Network-level functional connectivity | Baseline, 4-weeks, and 12 months
  The functional connectivity measure is derived from fMRI data acquired during a 10 minute period when the participant is in a state of wakefulness but has no directed task. In the analyses, fluctuations in activity within the Salience, Default Mode, and Looming networks throughout this period are correlated against other networks and regions to produce a measure of connectivity strength.
Network-level functional activation during fear conditioning | Baseline, 4-weeks, and 12 months
  Neural responses during fear conditioning are derived from fMRI data acquired when the participant is presented with faces, some of which have been associated with an aversive stimulus. In the analyses, activation within the Salience, Default Mode, and Looming networks during blocks of non-aversive and aversive stimulus presentations are directly contrasted to produce a measure of fear conditioning activation.
Looming network functional activation during fMRI looming paradigm | Baseline, 4-weeks, and 12 months
  Neural responses to looming stimuli are derived from fMRI data acquired when the participant is presented with faces which appear to move towards (approach) or away (withdraw) from the participant. In the analyses, Looming network activation during blocks of approaching face and withdrawing face presentations are directly contrasted to produce a measure of looming activation.
Arterial Spin Labeling -measured perfusion of the hippocampus and other regions | Baseline, 4-weeks, and 12 months
  Arterial Spin Labeling (ASL) fMRI data are acquired to assess cerebral blood flow (perfusion) within the hippocampus and other subcortical and cortical regions.
Neuromelanin-sensitive Magnetic Resonance Imaging in the midbrain | Baseline, 4-weeks, and 12 months
  Neuromelanin-sensitive Magnetic Resonance Imaging (NM-MRI) is a brain MRI technique capable of measuring MR signal intensity associated with neuromelanin (NM), a by-product of dopamine turnover, concentrated in the catecholamine-containing areas of the midbrain.
Structural Connectivity: Diffusion Tensor Imaging | Baseline, 4-weeks, and 12 months
  Diffusion Tensor Imaging (DTI) neuroimaging data are acquired to assess the structural connectivity between and within brain areas using the following metrics: Mean Diffusivity (MD), Axial Diffusivity (AD), Fractional anisotropy (FA), and Radial Diffusivity (RD).
Grade Point Average | Baseline, 12 months, and 24 months
  Each participant's grade point average (GPA) will be obtained from the academic registrar for each semester, as well as the cumulative GPA.
Registrar Enrollment Status Report | Baseline, 12 months, and 24 months
  The registrar enrollment status report will be obtained from the academic registrar, including records of any leaves of absence or withdrawals from college. The report will consist of categorical data indicating enrollment status as either: full-time (full course load), part-time (half course load), graduated, withdrawn (dropped out), or on leave (medical).
Health Services Utilization | Baseline, 12 months, and 24 months
  Health services utilization history will be obtained from the student health center reporting the frequency of on-campus behavioral health visits.
Mini-International Neuropsychiatric Interview - DSM 5 | Baseline, 4-weeks, 6 month, 12 months, and 24 months
  The Mini-International Neuropsychiatric Interview (MINI) - DSM 5 is a structured diagnostic interview to assess psychiatric diagnoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are sharing the data collected in this project via a two-tiered process via the NIMH Data Archive (http://nda.nih.gov/, NDA). The first tier is for the submission of descriptive/raw data while the study is ongoing. The second tier is for the submission of analyzed data at the time of the publication of results or when the study's primary aims have been achieved.
Supporting Information: CSR, Analytic Code
Time Frame: Study data will be come available once manuscripts are published.
Access Criteria: Data shared will be coded, with no PHI included.
URL: https://nda.nih.gov